CLINICAL TRIAL: NCT03000660
Title: A Phase I Trial of Venetoclax (ABT-199) and Dexamethasone for Relapsed or Refractory Systemic AL Amyloidosis
Brief Title: Trial of Venetoclax (ABT-199) and Dexamethasone for Relapsed or Refractory Systemic AL Amyloidosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: partial clinical hold per FDA
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AbbVie ABT-199
Record Dates: First submitted 2016-12-12; First posted 2016-12-22 (Estimated); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: AL Amyloidosis
Keywords: Amyloidosis; AL Amyloidosis; Amyloid Light Chain Amylodosis; ABT-199; Venetoclax
MeSH Terms: conditions — Immunoglobulin Light-chain Amyloidosis; Amyloidosis | interventions — venetoclax; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | US Export: No

ARMS (1):
- Venetoclax and Dexamethasone (Experimental): Venetoclax will be given at one of four escalating doses (100 mg/day, 200 mg/day, 400 mg/day, or 800 mg/day) by mouth on each day of the cycle. Dexamethasone will be given at 20mg by mouth on days 1, 8, 15, and 22 of each cycle.
  Interventions: Drug: Venetoclax; Drug: Dexamethasone

INTERVENTIONS:
Drug: Venetoclax — Venetoclax at one of four escalating doses
  Other Names: ABT-199
Drug: Dexamethasone — Dexamethasone 20mg by mouth on days 1, 8, 15, and 22 of each cycle.
  Other Names: Ozurdex; Maxidex; Baycadron

SUMMARY:
This is a study to determine the safety, tolerability and maximum tolerated dose of Venetoclax (ABT-199) and dexamethasone in relapsed or refractory amyloid light chain (AL) amyloidosis patients.

DETAILED DESCRIPTION:
The study is being conducted to determine the safety, tolerability and maximum tolerated dose of Venetoclax and dexamethasone in relapsed or refractory amyloid light chain (AL) amyloidosis patients. AL amyloidosis is a disease involving cells called plasma cells that make antibodies as part of your immune system. These cells are not functioning the way they are supposed to and they start to produce abnormal fragments of antibodies that are toxic to your body and can form amyloid. The antibody fragments are called "light chains." They can cause damage to organs, especially the kidneys, heart, skin, liver, and lungs.

Researchers are looking for ways to stop the light chains from being formed to treat the disease. Under some circumstances, patients will receive chemotherapy drugs in order to manage the disease. However, researchers do not know what the best treatment is for relapsed AL amyloidosis, so the researchers are testing new drugs or new combinations of drugs to see what will work best with the least side effects.

The researchers want to find out if Venetoclax (ABT-199) in addition to dexamethasone will reduce or eliminate AL amyloidosis plasma cells. In this study, varying doses of Venetoclax will be given to determine the maximum tolerated and safe dose for further study. The researchers may also gain a better understanding of whether Venetoclax and dexamethasone can counter the plasma cell disease that causes AL amyloidosis.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of AL amyloidosis, confirmed by positive Congo red stained biopsy, with evidence of measurable clonal disease according that requires active treatment
* Eastern Cooperative Oncology Group (ECOG) status of 0 to 2
* Relapsed or refractory after at least 1 prior therapy for AL amyloidosis and, in the investigator's opinion, require further treatment. Participants with a history of autologous stem cell transplantation must have adequate blood counts independent of growth factor support and have recovered from any transplant-related toxicities and be at least 100 days post-autologous transplant.
* Less than 30% plasma cells in the bone marrow biopsy and no bone lesions or hypercalcemia.
* The pre-screening test of CD138+ patient marrow plasma cells must show that the patient's CD138+ plasma cells have an apoptosis ratio of Venetoclax treated over untreated cells of greater than 1.4.
* Objective, measurable organ involvement. Skin purpura, carpal tunnel syndrome, or the presence of vascular amyloid on a bone marrow biopsy alone are not sufficient to meet criteria for "symptomatic organ involvement". Patients may have any of the following amyloid-related organ involvement as defined below:

  1. Renal: albuminuria higher than 0.5 g/day in a 24-hour urine collection.
  2. Cardiac: involvement is defined as the presence of a mean left ventricular wall thickness on echocardiogram more than 12 mm in the absence of a history of hypertension or valvular heart disease, or unexplained low voltage (< 0.5 mV) on electrocardiogram; or an NT-proBNP > 332 ng/L in CKD 1 or 2 patients or a BNP > 100ng/L in those who are CKD3.
  3. Hepatic: hepatomegaly on physical examination with alkaline phosphatase > 1.5 X the upper limit of normal (ULN).
  4. Autonomic or peripheral neuropathy: based on clinical history, autonomic dysfunction with orthostasis, symptoms of nausea or dysgeusia, gastric atony by gastric emptying scan, diarrhea or constipation, or abnormal sensory and/or motor findings on neurologic examination.
* AL Amyloidosis Cardiac Risk stage I, II or IIIa disease. Staging system defined by: NT-proBNP cut off of < 332 pg/mL and troponin I cut-off of < 0.10 ng/mL as thresholds for stages I, II and III; NT-proBNP < 8500 for stage IIIa.

  1. Stage I, both under threshold;
  2. Stage II, either troponin or NT-proBNP [but not both] over threshold;
  3. Stage III, both over threshold;
  4. Stage IIIa, both over threshold but NT-proBNP < 8500 pg/ml.
* Clinical laboratory values as specified below before the first dose of study drug:

  1. Echocardiographic ejection fraction > 45% within 28 days before the first dose of study drug.
  2. Within the 3 days of the first dose of study drug: i. Platelet count > 75 x 109/L; ii. Neutrophil count > 1.0 x 109/L; iii. Total bilirubin < 2 x ULN; iv. Alkaline phosphatase < 5 x ULN; v. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3 x ULN; vi. eGFR > 30 mL/min/1.73 m2
* Female patients who are postmenopausal for at least 1 year before the screening visit, OR are surgically sterile, OR, if they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 30 days after the last dose of study drug, or agree to completely abstain from heterosexual intercourse.
* Male patients, even if surgically sterilized (ie, status post vasectomy), who agree to practice effective barrier contraception during the entire study treatment period and through 30 days after the last dose of study drug, OR agree to completely abstain from heterosexual intercourse.
* Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.

Exclusion Criteria:

* Treatment with any investigational products within 28 days before the first dose of study drug.
* Requirement for other concomitant chemotherapy, immunotherapy, radiotherapy, or any ancillary therapy considered to be investigational.
* Failure to have fully recovered (ie, > Grade 1 toxicity) from the effects of prior chemotherapy regardless of the interval since last treatment.
* Active fungal infection requiring continued therapy.
* Cardiac system:

  1. QTc > 470 milliseconds (msec) on a 12 lead ECG obtained during the Screening period. If a machine reading is above this value, the ECG should be reviewed by a qualified reader and confirmed on a subsequent ECG.
  2. AL Amyloidosis Risk Stage IIIb disease. Stage IIIb is defined by NT-proBNP > 8500 pg/mL and troponin I > 0.10 ng/mL.
  3. New York Heart Association (NYHA) classification III or IV.
  4. Enzyme-documented myocardial infarction within 6 months before enrollment.
  5. Chronic atrial fibrillation.
  6. Grade 2 or 3 atrioventricular (AV) block (Mobitz, Type I permitted).
  7. Supine systolic blood pressure < 90 mmHg, or symptomatic orthostatic hypotension, or a decrease in systolic blood pressure on standing of > 20 mm Hg in spite of being treated for orthostatic hypotension.
  8. History of a bleeding diathesis or currently receiving treatment with warfarin. Patients are allowed to take aspirin.
* GI system:

  1. Severe diarrhea (= Grade 3) not controllable with medication (such as octreotide) or requires administration of total parenteral nutrition.
  2. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of study drug, including difficulty swallowing.
* Neurologic/ Social system:

  1. Patients with > Grade 2 peripheral neuropathy or painful peripheral neuropathy on clinical examination will be excluded.
  2. Previous or ongoing psychiatric illness.
  3. Social situations that would limit compliance with study requirements.
* Systemic infections:

  1. Known to be human immunodeficiency virus (HIV)-positive.
  2. Known to be hepatitis B surface antigen-positive or has known active hepatitis C infection.
  3. Uncontrolled infection requiring systemic antibiotics.
* Clinically overt multiple myeloma (bone marrow plasma cells > 30%) and bone lesions or hypercalcemia.
* Patients with non-AL amyloidosis.
* Presence of uncontrolled autoimmune hemolytic anemia or thrombocytopenia, or of active malignancy with the exception of non-melanoma skin cancer, cervical cancer, treated early-stage prostate cancer provided that prostate-specific antigen is within normal limit, or any completely resected carcinoma in situ.
* Female patients who are lactating or pregnant.
* Major surgery within 14 days before the first dose of study drug.
* Patients who are taking and are required to take any of the following agents that are CYP3A inhibitors: Amiodarone, Erythromycin, Fluconazole, Itraconazole, Ketoconazole, Miconazole, Diltiazem, Verapamil, Amprenavir, Fosamprenavir, Clarithromycin, Telithromycin, Nefazodone, Atazanavir, Darunavir, Indinavir, Lopinavir, Nelfinavir, Ritonavir, Saquinavir, Tipranavir.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-01; Primary Completion 2019-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Participants with treatment related adverse events using NCI CTCAE version 4.03. | Up to 8 months after beginning study drug
  Dose limiting toxicity will be based on hematologic and non-hematologic adverse events that are considered by the investigator to be possibly related to Venetoclax include any Grade 4 thrombocytopenia lasting more than 7 days, any Grade 4 neutropenia lasting more than 7 days, any Grade 3 or higher nonhematologic toxicity, a delay of more than 2 weeks in the initiation of Cycle 2 of treatment because of a lack of adequate recovery of Venetoclax-related hematological or nonhematologic toxicities, and any other Venetoclax-related nonhematologic toxicities Grade 2 or greater than, in the opinion of the investigator, requires discontinuation of therapy with Venetoclax. Also, events of concern that may be related to Venetoclax therapy will include worsening neuropathy, ventricular or atrial arrhythmia with hemodynamic instability, fluid retention that does not resolve with 3 or 4 days of intravenous diuretic therapy and bedrest, symptomatic congestive heart failure, and hypotension.

SECONDARY OUTCOMES:
Hematologic response based on serum free light chain (FLC) response criteria. | Up to 8 months after beginning study drug
  Complete response is normalization of FLC levels and ratio with negative immunofixation studies of serum and urine. Very good partial response is reduction of the difference between the involved and uninvolved FLC to less than 40mg/L. Partial response is reduction of the difference between involved and uninvolved FLC of greater than 50% baseline. No response or stable disease is none of the above.
Proportion of subjects with progression-free survival | Until disease progression up to three (3) years
  Hematologic progression will be evaluated every 12 weeks until the subject progresses. From CR any detectable monoclonal protein or abnormal free light chain ratio (light chain must double). From PR, 50% increase in serum M-protein of > 0.5 g/dl or 50% increase in urine M-protein to > 200 mg/day (a visible peak must be present), or free light chain increase of 50% to > 100 mg/L
Overall survival of subjects | From time of end of treatment to death for up to three (3) years
  Subjects will be followed until death after they have come off study

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Comenzo, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No